CLINICAL TRIAL: NCT01168154
Title: Phase 3 Study of Lactobacillus Reuterii in Patients With Symptomatic Non-complicated Diverticular Disease
Brief Title: Role Of Lactobacillus Reuteri DSM 17938 In The Non-Complicated Diverticular Disease
Acronym: ReDiCo
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Collaborators: Careggi Hospital (Other)
Responsible Party: Fabrizio Bossa, Casa Sollievo della Sofferenza Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ReDiCo
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2008-10

CONDITIONS: Diverticulosis; Diverticulitis
Keywords: Diverticula; Diverticular disease; Diverticulitis; Probiotics
MeSH Terms: conditions — Diverticulum; Diverticulitis; Diverticular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus Reuterii (Active Comparator)
  Interventions: Dietary Supplement: Lactobacillus Reuterii
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus Reuterii — Lactobacillus Reuterii 10000000000 CFU per day
  Arms: Lactobacillus Reuterii
Dietary Supplement: placebo — placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effectiveness and the tolerability of the Lactobacillus reuteri in the control of the diverticular disease symptoms and in the prevention of acute diverticulitis episodes.

DETAILED DESCRIPTION:
The gastrointestinal apparatus hosts a bacterial population that quantifies to around 1011 microorganisms per gram of content with more than 400 different species. Its principal functions are: metabolic, trophic, and protective. The Lactobacillus reuteri (Reuterin®) is considered one of the few native species in the human intestinal tract. It is able to modulate the immune response CD4+ T-Helper to an ileum level. Lactobacillus reuteri isolated for the first time in 1980 is a heterofermantative species. Its probiotic activity is attributed to the ability to exercise an inhibitive effect on the pathogenic micro-organisms with a combination of mechanisms including the production of lactic acid, hydrogen peroxide, antimicrobic substances and bactericide. Moreover, Lactobacillus reuteri is in a position to produce various short chain-like fat acids such as the acetic acid from the fermentation of carbohydrates. At last, it is in a position to produce a powerful antimicrob substance known as Reuterina that is capable of inhibiting the growth of many bacterial species including Escherichia, Salmonella, Shigella, Proteus, Pseudomonas, Clostridium and Sfafilococcus as well as fungi and protozoa, many of which are pathogens for man.

Among pathologies in which it is hypothesized that probiotics could have a possible therapeutic role, there is the diverticulosis disease. Approximately 20% of patients with colonic diverticula have intestinal disturbances and a reduction of the quality of life. Moreover approximately 20% of the patients with diverticulosis in the colon have at least 1 acute diverticulitis attack, characterized by pain, fever, abdominal defence, increment of the VES and neutrophil leucocytosis. Usually the acute diverticulitis episode can be controlled by medical therapy, but repeated episodes in time often lead to greater complications in the perforation, from the abdominal abscesses, from the fistulas and from the stenosis. The prevention of acute diverticulitis episodes is therefore very important so as to prevent greater complications of such pathology.

Until now, the scientific evidences have suggested the use of fibre and non-absorbable antibiotics (such as rifaximine) for the treatment of a non-complicated diverticular disease and for the prophylaxis of the feared complications. The extended use of antibiotics exposes to the risk of selecting resistant strains and there are no long-term studies on the outcome of the patients suffering from diverticulosis in continuous therapy with rifaximine and fibres. The therapy with Lactobacillus reuteri could be effective in the control of symptoms of the diverticular disease through its trophic action on coloncytes (thanks to the SCFA production), both through the modulation of the activity of the immune system and on the intestinal permeability. Moreover the antibacterial activity of Lactobacillus reuteri against the pathogenic bacteria could be useful in the prevention and the treatment of acute diverticulitis episodes. Finally, thanks to its trophic role on the intestinal epithelium, Lactobacillus reuteri could help the mucosal cure of acute diverticulitis episodes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients affected by symptomatic diverticulosis
* Informed consent obtained and signed.
* Expected compliance

Exclusion Criteria:

* Patients supplemented with other probiotics
* Patients treated with antibiotics
* Patients affected by hearth failure, renal failure, neoplasia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of 50% of the score of activity of the diverticular disease | 1 year
  A validated questionnaire was used to investigate on intestinal symptoms. The following symptoms/signs will be investigated:
  * Abdominal pain
  * Abdominal bloating
  * Urgency
  * Diarrhoea
  * Abdominal Tension
  Each factor previously listed will be graded according to the following scale of gravity:
  * 0= no symptom
  * 1= light disturbance
  * 2= moderate disturbance
  * 3= serious disturbance The score of activities can range between 0 (asymptomatic patient) to 15 (serious disturbances with important impacts on the quality of life).

SECONDARY OUTCOMES:
Reduction of 20% of acute diverticulitis episodes | 1 year
  To value the efficancy in reduction of acute diverticulitis, defined as episodes of abdominal pain associated with fever and/or abdominal resistance, increment of ESR and neutrophil leucocitosis and that demand a treatment of systemic antibiotics

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Careggi Hospital, Florence
  - Casa Sollievo della Sofferenza Hospital - IRCCS, San Giovanni Rotondo